CLINICAL TRIAL: NCT03408535
Title: Assessing the Feasibility of a Clinical Trial of an Online Audiological Rehabilitation Program
Brief Title: Feasibility of an Online Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Eriksholm Research Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RGS 16086; IRAS Project id: 214225 (Other: National Health Service Health Research Authority); 16IH008 (Other: Nottingham University Hospitals NHS Trust)
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
Keywords: eHealth; Online Rehabilitation; Hearing Problems; Adult; Hearing Aids
MeSH Terms: conditions — Hearing Loss; Hearing Disorders

STUDY DESIGN:
Intervention Model Description: A single-centre feasibility study of a clinical study with one arm (intervention-only). A before and after intervention design will be used. A sub-group of participants will take part in a qualitative follow-up session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eriksholm Guide to Better Hearing (Other): The Eriksholm Guide to Better Hearing is an online rehabilitation program. The program is made up of 5-weekly modules that cover different topics. Each module includes self-studies, training, and professional video coaching in hearing loss, hearing aids, and communication strategies.
  Interventions: Other: Eriksholm Guide to Better Hearing

INTERVENTIONS:
Other: Eriksholm Guide to Better Hearing — Online rehabilitation program.

SUMMARY:
The study will assess the feasibility of conducting a full-scale clinical trial of the effectiveness of an online rehabilitation program for adults living with hearing loss. The program aims to help people use their hearing aid(s) and interact in social settings more effectively. The program is made up of 5 modules that cover different topics, such as hearing aids, communication strategies, and relaxation techniques.

DETAILED DESCRIPTION:
STUDY PURPOSE

This feasibility study is a precursor of a randomised controlled trial (RCT) that will evaluate the effectiveness of an English-speaking version of the online program originally evaluated by Thorén et al in adult hearing aid users. This study will estimate a number of parameters necessary for the robust design of an RCT. This systematic approach of completing a feasibility study prior to a full-scale evaluation is strongly advocated by the Medical Research Council (MRC) guidelines for developing and evaluating complex interventions, ensuring that any uncertainties are addressed and that the intervention operates as intended.

OBJECTIVES

This study will be used to estimate the following parameters:

(I) Recruitment

1. Willingness of clinicians to recruit participants
2. Willingness of participants to consent
3. Number of eligible patients.

(II) Feasibility/acceptability of approach (Quantitative outcomes)

1. Characteristics of the outcome measures
2. Standard deviation of outcome measures to estimate sample size
3. Follow-up rates, response rates to questionnaires, adherence/compliance rates
4. Time needed to collect and analyse data.

(III) Users' perspective/opinions of the intervention (Qualitative outcomes)

1. Participant's views regarding delivery of the program through different devices
2. How the program is used and how often (i.e. usability)
3. Participants views concerning what they like and dislike about the program (i.e.

   acceptability)
4. How much of the program is completed (adherence).

STUDY CONFIGURATION

A single-centre feasibility study of a clinical study with one arm (intervention-only). A before and after intervention design will be used. A sub-group of participants will take part in a qualitative follow-up session.

Primary endpoint. In accordance with objective (II) feasibility/acceptability of approach, follow-up measures will be recorded upon completion of the last intervention module

Secondary endpoint. In accordance with objective (III) users' perspective/opinions of the intervention, completion of focus groups.

Participant Duration. Participants will take part in an initial assessment, which is estimated to last 1.5 hours. After completing the weekly online modules from home, participants will then take part in a follow-up assessment which will last up to 1.5 hours. A sub-sample of 16 participants will also be invited to take part focus groups lasting 1.5 hours (end of the study).

Recruitment. Existing hearing aid users will be identified from the National Institute for Health Research (NIHR) Nottingham Biomedical Research Centre (BRC) Otology and Hearing Group's participant database. Participants in this database have provided consent to be approached about future research studies.

First-time hearing aid users will be recruited from publically funded National Health Service (NHS) Adult Audiology Departments in the East Midlands, UK.

All participants who express an interest in the study will receive a participant information sheet, alongside a pre-paid, addressed envelope in which to return their response if they choose to take part.

STATISTICS

Methods. The study data will be analysed by the research team at the NIHR Nottingham BRC. All data will be analysed on University of Nottingham computers and backed up to the University of Nottingham servers. Data will be analysed using STATA version 14. Continuous data will be summarised using means and standard deviations, whereas categorical data will be summarised using percentages. For each measure, the difference between baseline and follow-up will be examined using a paired samples t-test or Wilcoxon signed rank test. Medians and quartiles will be reported for non-parametric data, and means, standard deviations and 95% confidence intervals for parametric data. Statistical significance will be set at p=.05. As outcome data will be collected after the intervention period, no interim analyses will be performed.

Sample size and justification. The sample size estimate is based on the difference between two dependent means; baseline and follow-up. An a priori sample size calculation (G*power v.3.0.10) based on a medium effect size (Cohen's d=0.5), a one-sided Type I error rate of 5%, and 80% power, revealed that a sample size of 27 participants will be required for each sample (first-time and existing hearing aid users).

Assessment of efficacy. This is a feasibility study of a clinical study and, as such, will not assess the efficacy of the online rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* English as first spoken language or good understanding of English.
* Adults aged ≥18 years (no upper age limit)
* Mild-to-moderate hearing loss (average hearing threshold across octave frequencies 0.25-4kHz ≥20 and ≤70dB HL)
* Have either:

  1. Used hearing aids for at least one year (existing hearing aid users), or
  2. Have not used hearing aids or an alternative form of amplification (e.g. personal sound amplification products) within the past two years (first-time hearing aid users)
* Access the Internet and compatible device (e.g. computer or tablet device).

Exclusion Criteria:

* Report having severe tinnitus
* Diagnosis of Ménière's disease
* Patients who are unable to complete the questionnaires without assistance due to age- related problems such as cognitive decline and dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE: Ventry & Weinstein, 1982) | Change from Baseline following up to 5 weeks of independent use of the online intervention
  A 25-item questionnaire designed to assess the effects of hearing loss on the emotional (n = 13), and social/situational adjustment (n = 12) of older people, scored using a three-point scale (4 = yes; 2 = sometimes; 0 = no).

SECONDARY OUTCOMES:
International Outcome Inventory for Hearing Aids (IOI-HA: Cox & Alexander, 2002) | Baseline and following up to 5 weeks of independent use of the online intervention
  A seven-item questionnaire (use, benefit, residual activity limitation, satisfaction, residual participation restriction, importance to others, quality of life) and is scored on a five-point scale.
Glasgow Hearing Aid Benefit Profile (GHABP: Gatehouse, 1999) | Baseline (Part 1 only) and following up to 5 weeks of independent use of the online intervention (Part 2 only)
  Assesses hearing disability (or activity limitations) and handicap (or participation restrictions; part 1), and hearing aid use, benefit, residual disability and satisfaction (part 2). Each domain is measured on a five-point scale.
Social Participation Restrictions Questionnaire (SPaRQ: Heffernan et al., 2016) | Baseline and following up to 5 weeks of independent use of the online intervention
  A 19-item inventory that assesses social behaviours (9-items) and perceptions (10-items) in adults with mild-to-moderate hearing loss. Each item is measured on an 11-point response scale ranging from 'Completely Disagree' at point zero to 'Completely Agree' at point ten.
Measure of Audiologic Rehabilitation Self-efficacy for Hearing Aids (MARS-HA: West & Smith, 2007) | Baseline and following up to 5 weeks of independent use of the online intervention
  Includes four subscales: basic handling, advanced handling, adjustment to hearing aids, and aided listening skills. Respondents indicate how confident they are that they could do the things described on an 11-point scale (0%=cannot do this, to 100%=certain I can do this).
Practical Hearing Aid Skills Test (PHAST: Desjardins & Doherty, 2009) | Baseline and following up to 5 weeks of independent use of the online intervention
  Tests eight hearing aid skills (insertion, removal, opening battery door, changing the battery, cleaning the aid, manipulating the voice clarity (VC), telephone use, and use of programs). Each skill was scored on a five-point Likert scale (0=cannot perform, 4=excellent).
Hearing Aid and Communication Knowledge (HACK: Ferguson et al, 2015) | Baseline and following up to 5 weeks of independent use of the online intervention
  A 20-item open-ended questionnaire that measures free recall of knowledge relevant to practical (n = 12) and psychosocial (n = 8) issues on hearing aids and communication.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Health Research (NIHR) Nottingham Biomedical Research Centre, Nottingham, Non-US/Non-Canadian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoren ES, Oberg M, Wanstrom G, Andersson G, Lunner T. A randomized controlled trial evaluating the effects of online rehabilitative intervention for adult hearing-aid users. Int J Audiol. 2014 Jul;53(7):452-61. doi: 10.3109/14992027.2014.892643. Epub 2014 Apr 22. PMID 24749664
- [Background] Thoren E, Svensson M, Tornqvist A, Andersson G, Carlbring P, Lunner T. Rehabilitative online education versus internet discussion group for hearing aid users: a randomized controlled trial. J Am Acad Audiol. 2011 May;22(5):274-85. doi: 10.3766/jaaa.22.5.4. PMID 21756843
- [Background] Ventry IM, Weinstein BE. The hearing handicap inventory for the elderly: a new tool. Ear Hear. 1982 May-Jun;3(3):128-34. doi: 10.1097/00003446-198205000-00006. PMID 7095321
- [Background] Cox RM, Alexander GC. The International Outcome Inventory for Hearing Aids (IOI-HA): psychometric properties of the English version. Int J Audiol. 2002 Jan;41(1):30-5. doi: 10.3109/14992020209101309. PMID 12467367
- [Background] Gatehouse S. Glasgow Hearing Aid Benefit Profile: Derivation and validation of client-centred outcome measures for hearing aid services. J Am Acad Audiol. 1999;10(2):80-103.
- [Background] Heffernan E, Coulson N, Henshaw H, Barry J, Ferguson MA. The development of a measure of participation in adults with hearing loss: a qualitative study of expert views. Trials. 2015;16(Suppl 1):30.
- [Background] West RL, Smith SL. Development of a hearing aid self-efficacy questionnaire. Int J Audiol. 2007 Dec;46(12):759-71. doi: 10.1080/14992020701545898. PMID 18049965
- [Background] Desjardins JL, Doherty KA. Do experienced hearing aid users know how to use their hearing AIDS correctly? Am J Audiol. 2009 Jun;18(1):69-76. doi: 10.1044/1059-0889(2009/08-0022). Epub 2009 Apr 20. PMID 19380509
- [Background] Ferguson M, Brandreth M, Brassington W, Wharrad H. Information Retention and Overload in First-Time Hearing Aid Users: An Interactive Multimedia Educational Solution. Am J Audiol. 2015 Sep;24(3):329-32. doi: 10.1044/2015_AJA-14-0088. PMID 26649541
- [Background] Medical Research Council. Developing and evaluating complex interventions: new guidance. 2006. Retrieved from: https://www.mrc.ac.uk/documents/pdf/complex-interventions-guidance/.